CLINICAL TRIAL: NCT04154865
Title: Exercise in Adolescents With Insulin Resistance: A Path to Improved Brain Health?
Brief Title: Exercise in Adolescents With Insulin Resistance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment failure
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-0838; 2019-0838 (Other: Institutional Review Board); A176000 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison); Protocol Version 2/10/2023 (Other: UW Madison)
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Ultrasonography, Doppler, Transcranial; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled, eligible (Experimental): Single arm for eligible subjects
  Interventions: Other: Hypercapnia; Device: Transcranial Doppler; Device: Cycle ergometer; Other: Cognitive Tests

INTERVENTIONS:
Other: Hypercapnia — Eligible subjects will undergo transcranial Doppler assessment before and after hypercapnia exposure.
  Other Names: CO2
Device: Transcranial Doppler — A transcranial Doppler ultrasound probe will be used to assess middle cerebral artery velocity to quantify cerebral blood flow at various time points throughout the study visit.
  Other Names: TCD
Device: Cycle ergometer — A cycle ergometer will be used to acutely increase cerebral blood flow.
  Other Names: Stationary bike
Other: Cognitive Tests — A battery of cognitive tests will be completed by the subject.

SUMMARY:
The growing population of adolescents with insulin resistance (IR) is predicted to create a large public health burden in the next few decades. This study examines the function of brain blood vessels and cognitive function, to test if increasing severity of IR in adolescents is related to reduced cognitive function and reduced brain blood vessel function. Findings from this study may help create treatments to delay or prevent some of the negative effects of IR on cognitive and vascular health.

DETAILED DESCRIPTION:
Insulin resistance (IR), a hallmark of metabolic syndrome and diabetes, is strongly linked to numerous health disorders, including cardiovascular and cerebrovascular disease. In adults, data indicate IR negatively impacts brain structure and function, such as decreased regional brain volumes, increased white matter hyperintensities, and poorer memory and attention, all of which are hallmarks of Alzheimer's disease and related dementias. In parallel with data from adults, emerging data from adolescents with IR suggest similar brain structural and functional changes. Importantly, these changes occur during a critical period for proper brain development and maturation, thus having a potentially fateful impact on these young brains as they mature into adulthood.

In addition to brain structural and cognitive changes, IR is also associated with lower cerebral blood flow (CBF), which is linked to neurocognitive problems in adults. The consequences of IR on cerebrovascular dysfunction- and its interaction with neurocognition- in adolescents remain largely unexplored. Therefore, impaired vascular function may hold tremendous influence over brain health in adolescents at a vital period in brain development.

Exercise is a key factor in treating IR from a metabolic perspective, and acts as the only effective intervention known to combat dementia-related diseases in adults. Furthermore, exercise can acutely increase cognitive abilities and CBF, and adults with higher aerobic fitness demonstrate greater CBF, and CBF is increased following exercise training. With this as background, a few questions emerge regarding adolescents with IR: is there a dose-response relationship between IR severity and cognitive function? Can exercise improve cognition and impact brain health? What is the role of vascular function in cognition on potential exercise-induced improvements?

The long-term goal of this research program is to determine the influence of IR, physical activity, and their interaction on brain development in adolescents by interrogating the relationships between neurocognition, brain structure, and underlying mechanisms. The primary goal of the current pilot project is to quantify neurocognitive function in relation to the severity of IR and use acute exercise as a tool to improve function. The central hypothesis is that as IR worsens: 1) subtle neurocognitive abnormalities worsen, 2) exercise-mediated improvements in neurocognitive function are blunted, due in part to 3) reduced CBF responses.

Participants will be recruited primarily from pediatric and pediatric endocrinology clinics via our collaborator, Dr. Aaron Carrel, and his staff in UWHC Pediatric Endocrinology. Additionally, participants will be recruited from the greater Madison, WI community.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18 years inclusive
* Typically developing and cognitively intact

Exclusion Criteria:

* Diabetes (≥126 mg dL-1 fasting glucose)
* Insulin treatment or sensitizing drugs
* Diagnosis of kidney, pulmonary, or heart disease (an asthma diagnosis that is not currently being treated with a daily controller medicine or asthma that requires medication use prior to exercise is not considered a pulmonary disease)
* Current smoking (defined as use of nicotine >5 times in the past month)
* Pregnancy
* Neurological or developmental disorders (e.g., intellectual disability, autism)
* Significant head injury or medical conditions (e.g., concussion, encephalopathy, seizure disorder)
* Inability to undergo the MRI procedure
* Weight less than 94.5 lbs (42.9 kg) to adhere to safety guidelines regarding blood sampling and OGTT administration
* Tanner Stage <3
* Any other circumstance deemed by the PI not addressed above

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Cognitive Function as determined by NIH Toolbox Picture Vocabulary Test | up to 1 day
  Participants will undergo a series of cognitive tests to evaluate intelligence, memory, speed function, executive function, and psychiatric quality of life. The results of these test will be scored and reported individually.
  The NIH Toolbox Picture Vocabulary Test assesses the mental processes that translate thought into symbols (words, gestures) that can be shared among individuals for purposes of communication. The respondent is presented with an audio recording of a word and four photographic images on the computer screen and is asked to select the picture that most closely matches the meaning of the word. This test is scored by the total number of correct responses with a total range of possible scores 0-130 with higher scores indicating better vocabulary skills.
Cognitive Function as determined by NIH Flanker Inhibitory Control and Attention Test | up to 1 day
  Participants will undergo a series of cognitive tests to evaluate intelligence, memory, speed function, executive function, and psychiatric quality of life. The results of these test will be scored and reported individually.
  The NIH Toolbox Flanker Inhibitory Control and Attention Test assess executive attention. It is a visual display using a central arrow flanked by arrows either pointing in the same direction or different that the central arrow. The participant is to indicate the direction of the central arrow when they are all pointing in the same direction. Scoring is algorithm derived and based on accuracy and reaction time, with a total range of possible scores 0-10 with higher scores indicating increased executive attention.
Cognitive Function as determined by NIH List Sorting Working Memory Test | up to 1 day
  Participants will undergo a series of cognitive tests to evaluate intelligence, memory, speed function, executive function, and psychiatric quality of life. The results of these test will be scored and reported individually.
  The NIH Toolbox List Sorting Working Memory Test assesses working memory by having participants sort images by size order. The total range of possible score is 0-28, with higher scores indicating more improved working memory.
Cognitive Function as determined by NIH Dimensional Change Card Sorting Test | up to 1 day
  Participants will undergo a series of cognitive tests to evaluate intelligence, memory, speed function, executive function, and psychiatric quality of life. The results of these test will be scored and reported individually.
  The NIH Dimensional Change Card Sorting Test assesses cognitive flexibility and attention. Two target pictures are presented that vary along two dimensions (e.g., shape and color). Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape). "Switch" trials are also employed, in which the participant must change the dimension being matched. Scoring is based on a combination of accuracy and reaction time with a total range of possible scores 0-10 with higher scores indicating increased cognitive flexibility and attention.
Cognitive Function as determined by NIH Pattern Comparison Test | up to 1 day
  Participants will undergo a series of cognitive tests to evaluate intelligence, memory, speed function, executive function, and psychiatric quality of life. The results of these test will be scored and reported individually.
  The NIH Toolbox (Pattern Completion) assesses processing speed by asking participants to indicate if visual stimuli are the same or not the same. This test is scored by the total number of correct responses in 90 seconds (maximum score is 130). The higher the score, the better the processing speed.
Cognitive Function as determined by NIH Picture Sequence Test | up to 1 day
  Participants will undergo a series of cognitive tests to evaluate intelligence, memory, speed function, executive function, and psychiatric quality of life. The results of these test will be scored and reported individually.
  The NIH Toolbox (Picture Sequence) assesses episodic memory. Participants are shown a series of pictures one at a time, related to a single theme. After the last picture is shown, the participants is asked to place the pictures in the demonstrated sequence. The total number of correct placements across 3 trials provides the score, up to a maximum of 48. The higher the score, the better the episodic memory.
Cognitive Function as determined by NIH Oral Reading Recognition Test | up to 1 day
  Participants will undergo a series of cognitive tests to evaluate intelligence, memory, speed function, executive function, and psychiatric quality of life. The results of these test will be scored and reported individually.
  The NIH Toolbox Oral Reading Recognition Test assesses reading decoding skill and of crystallized abilities. The participant is asked to read and pronounce letters and words as accurately as possible. Scoring is based on the number of correct items with a possible score up to 2500. The higher the score, the better the crystallized abilities.
Cognitive Function as determined by PedsQL - (Child 8-12/Teen 13-18) | up to 1 day
  Participants will undergo a series of cognitive tests to evaluate intelligence, memory, speed function, executive function, and psychiatric quality of life. The results of these test will be scored and reported individually.
  The Pediatric Quality of Life Inventory (PedsQL) is a 23-item survey assessing 4 functional dimensions: Physical, Emotional, Social, and School. Each item is scored on a 5-point Likert scale where 0 is 'not at all' and 4 is 'almost always'. Items are reversed scored (0=100, 1=75, 2=50, 3=25, 4=0) and linearly transformed to a 1-100 scale, where the higher the score, the better the Quality of Life.
Cerebral blood flow as determined by TCD | up to 1 day
  CBF will be measured via TCD before (baseline) and after CO2 at 6 minutes; and before (baseline) and during exercise at 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: William Schrage, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04154865/ICF_000.pdf